CLINICAL TRIAL: NCT00673569
Title: A Phase II Single-Arm Trial Assessing the Use of an Ex Vivo Sensitivity Assay to Predict Response of Relapsed Metastatic Non-Small Cell Lung Cancer Patients to Erlotinib
Brief Title: Laboratory Test in Predicting Response to Erlotinib in Patients With Relapsed Metastatic or Unresectable Non-Small Cell Lung Cancer That Did Not Respond to Previous Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Charles M. Rudin, Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Masking: None | Purpose: Treatment
Other Study IDs: JHOC-J0655, CDR0000512886; P30CA006973 (NIH); JHOC-J0655
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2010-08

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IV non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Gene Expression Profiling; Immunoenzyme Techniques; Immunologic Techniques; Biopsy, Needle

INTERVENTIONS:
Drug: erlotinib hydrochloride
Genetic: gene expression analysis
Genetic: protein expression analysis
Other: immunoenzyme technique
Other: immunologic technique
Other: laboratory biomarker analysis
Procedure: needle biopsy

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer. It may also help doctors learn how well patients will respond to treatment.

PURPOSE: This phase II trial is studying how well a laboratory test predicts response to erlotinib in patients with metastatic or unresectable non-small cell lung cancer that did not respond to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether the extent of inhibition of ERK phosphorylation in lung cancer cells exposed ex vivo and in vivo to erlotinib hydrochloride significantly differs between responding and nonresponding patients with relapsed, metastatic or unresectable non-small cell lung cancer.

Secondary

* Determine whether the extent of inhibition of epidermal growth factor receptor (EGFR) and AKT phosphorylation in lung cancer cells exposed ex vivo and in vivo to erlotinib hydrochloride significantly differs between these 2 groups of patients.
* Correlate the extent of inhibition of EGFR, ERK, and AKT phosphorylation in lung cancer cells exposed ex vivo with erlotinib hydrochloride with in vivo objective tumor response to erlotinib hydrochloride in these patients.
* Correlate EGFR gene mutation and amplification status with pharmacodynamic evidence of response to erlotinib hydrochloride in these patients.

OUTLINE: This is an open-label, pilot study.

Patients receive oral erlotinib hydrochloride once daily on days 1-28. Treatment repeats every 28 days for at least 2 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo tumor fine-needle aspiration biopsies under ultrasound or CT scan guidance at baseline and between days 12-15 for laboratory studies. Laboratory studies include quantitative western blot and enzyme-linked immunosorbent assays, gene mutation and amplification, and ex vivo assays. Tumor cells are also analyzed for changes in phosphorylation status and/or expression levels of pharmacodynamic markers, including total- and phospho-epidermal growth factor receptor, total- and phospho-ERK, and total- and phospho-AKT.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic or unresectable non-small cell lung cancer
* Relapsed disease

  * Failed ≥ 1 prior chemotherapy regimen
* Measurable disease
* Tumor must be accessible to fine-needle aspiration
* No uncontrolled brain metastases

  * Patients with brain metastases must have stable neurologic status after local therapy (surgery or radiotherapy) for ≥ 4 weeks and no neurologic dysfunction that would preclude evaluation of neurologic and other adverse events

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 12 weeks
* WBC > 3,000/mm³
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 100,000/mm³
* Bilirubin normal
* PT and activated PTT normal
* Creatinine normal OR creatinine clearance > 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled intercurrent illness, including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would preclude study compliance
* No significant ophthalmologic abnormalities*, including any of the following:

  * Severe dry eye syndrome
  * Keratoconjunctivitis sicca
  * Sjögren's syndrome
  * Severe exposure keratopathy
  * Disorders that might increase the risk for epithelium-related complications (e.g., bullous keratopathy, aniridia, severe chemical burns, or neutrophilic keratitis)
* No serious, nonhealing wound, ulcer, or bone fracture
* No significant traumatic injury within the past 14 days NOTE: *Patients with mild forms of any of the above ophthalmologic abnormalities, an asymptomatic history, or a normal ophthalmologic examination allowed at the discretion of the investigator. Patients with treatable conditions (e.g., infectious keratitis/conjunctivitis or allergic conjunctivitis) allowed after treatment or resolution of the condition.

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior small molecule inhibitors of epidermal growth factor receptor, including erlotinib hydrochloride or gefitinib
* At least 4 weeks since prior anticancer therapy, including chemotherapy, radiotherapy, biologic therapy, or other investigational therapy (6 weeks for nitrosoureas or mitomycin C)
* More than 14 days since prior major surgery or open biopsy and recovered
* At least 7 days since prior and no concurrent inhibitors of CYP3A4, including any of the following:

  * Itraconazole
  * Herbal extracts and tinctures, including any of the following:

    * Hydrastis canadensis (goldenseal)
    * Uncaria tomentosa (cat's claw)
    * Echinacea angustifolia roots
    * Trifolium pratense (wild cherry)
    * Chamomile
    * Licorice root
    * Dillapiol
    * Naringenin
* No concurrent inducers of CYP3A4, including any of the following:

  * Phenytoin
  * Carbamazepine
  * Rifampin
  * Barbiturates
  * Hypericum perforatum (St. John's wort)
* No concurrent chemotherapy
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent radiotherapy, including palliative radiotherapy
* No concurrent therapeutic anticoagulation
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-09; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Quantitative assessment of phospho-ERK
Extent of inhibition of ERK phosphorylation by erlotinib hydrochloride
Clinical response

SECONDARY OUTCOMES:
Extent of inhibition of epidermal growth factor receptor (EGFR) and AKT phosphorylation by erlotinib hydrochloride
Toxicity
Frequency and proportion of patients with complete response, partial response, stable disease, and progressive disease
Comparison of ex vivo and in vivo effects of erlotinib hydrochloride
Proportion of patients with EGFR gene amplification and gene mutation with an ex vivo response and clinical response

CONTACTS AND LOCATIONS:
Overall Officials: Charles M. Rudin, MD, PhD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States